CLINICAL TRIAL: NCT01203241
Title: Benefit of Left Atrial Roof Ablation in Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, Head of the Arrhythmia Unit, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LARA-PAF
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Drug-refractory Paroxysmal Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Conventional ablation (Active Comparator): Pulmonary vein encircling by performing continuous radiofrequency lesions surrounding each ipsilateral pulmonary vein antrum
  Interventions: Procedure: Pulmonary vein encircling
- Conventional ablation plus left atrial roof ablation (Active Comparator): Pulmonary vein encircling by performing continuous radiofrequency lesions surrounding each ipsilateral pulmonary vein antrum plus creation of a radiofrequency line joining contralateral superior pulmonary veins throughout the left atrial roof.
  Interventions: Procedure: Pulmonary vein encircling plus roof ablation

INTERVENTIONS:
Procedure: Pulmonary vein encircling — Pulmonary vein encircling by performing continuous radiofrequency lesions surrounding each ipsilateral pulmonary vein antrum
  Arms: Conventional ablation
Procedure: Pulmonary vein encircling plus roof ablation — Pulmonary vein encircling by performing continuous radiofrequency lesions surrounding each ipsilateral pulmonary vein antrum plus creation of a radiofrequency line joining contralateral superior pulmonary veins throughout the left atrial roof.
  Arms: Conventional ablation plus left atrial roof ablation

SUMMARY:
The aim of the present study is to assess whether left atrial roof ablation adds any benefit in the arrhythmia-free probability after paroxysmal atrial fibrillation ablation.

ELIGIBILITY:
Inclusion Criteria:

* Drug-refractory paroxysmal atrial fibrillation

Exclusion Criteria:

* Hypo or hyperthyroidism
* Implantable defibrillation or pacemaker implanted
* Moderate or severe mitral valve disease or mitral prosthetic valve
* Ejection fraction less than 30%
* Left atrial anteroposterior diameter more than 50 mm.
* Previous atrial fibrillation ablation
* Left atrium thrombus
* Current infective disease or sepsis
* Pregnant women
* Current unstable angor
* Acute myocardial infarction in last 3 months
* Atrial fibrillation secondary to ionic disturbance, thyroids disease or secondary to any other reversible or non cardiovascular disease
* Reduced expectancy of life (less than 12 months)
* Patient participating in another clinical study that investigates a drug or device
* Psychologically unstable patient or denies to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial arrhythmias without antiarrhythmic drugs | 1-year follow-up

SECONDARY OUTCOMES:
Freedom from atrial arrhythmias with or without antiarrhythmic drugs | 1-year follow-up
Presence of any complications in the acute phase or during follow-up | 1-year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic Universitari, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Arbelo E, Guiu E, Ramos P, Bisbal F, Borras R, Andreu D, Tolosana JM, Berruezo A, Brugada J, Mont L. Benefit of left atrial roof linear ablation in paroxysmal atrial fibrillation: a prospective, randomized study. J Am Heart Assoc. 2014 Sep 5;3(5):e000877. doi: 10.1161/JAHA.114.000877. PMID 25193295